CLINICAL TRIAL: NCT07061756
Title: Characteristics of Subgingival Microbiota in Patients With Stage III-IV Periodontitis in Response to Nd:YAG Laser-Assisted Therapy
Brief Title: Nd:YAG Laser Effects on Subgingival Microbiota in Stage III-IV Periodontitis
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rui He (Other)
Responsible Party: Sponsor-Investigator, Rui He, Resident Physician, First Affiliated Hospital, Sun Yat-Sen University
Organization: First Affiliated Hospital, Sun Yat-Sen University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: [2024]493-1
Record Dates: First submitted 2025-06-19; First posted 2025-07-11 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-06

CONDITIONS: Periodontitis
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nd group (Experimental): The Nd group received comprehensive periodontal therapy combining scaling and root planing (SRP) with adjunctive Nd:YAG laser treatment.
  Interventions: Procedure: ND
- SRP group (Active Comparator): The SRP group received standard periodontal therapy consisting of scaling and root planing (SRP) alone, serving as the active control for comparison against laser-assisted treatment.
  Interventions: Procedure: SRP

INTERVENTIONS:
Procedure: SRP — Full-mouth scaling and root planing (SRP) was performed using an ultrasonic scaler (EMS AIR-FLOW MASTER PIEZON®) supplemented by Gracey curettes for subgingival instrumentation. All procedures were conducted under local anesthesia by a calibrated periodontist, with each quadrant treated for a minimum of 30 minutes. Patients received standardized oral hygiene instructions and were scheduled for a 3-month postoperative follow-up.
  Arms: SRP group
Procedure: ND — In addition to the identical SRP protocol described above, adjunctive Nd:YAG laser therapy (Wiser Waterlase MD, Vista Dental) was applied immediately post-SRP. Laser parameters were set at 150 mJ/pulse, 20 Hz frequency with water (level 1) and air (level 3) coolant. The fiber optic tip (300 μm diameter) was moved in a continuous "Zig-zag" pattern along the root surface and pocket epithelium, maintaining 2-second irradiation per site at a 30° angle to the tooth axis. Standardized oral hygiene instructions and 3-month follow-up were similarly provided.
  Arms: Nd group

SUMMARY:
This randomized controlled trial (RCT) aims to evaluate the clinical efficacy of Nd:YAG laser adjunctive therapy and its impact on the subgingival microbiome in patients with stage III-IV periodontitis. The study addresses two key questions: (1) Whether Nd:YAG laser combined with scaling and root planing (SRP) yields significantly greater improvements in periodontal parameters compared to SRP alone; and (2) How subgingival microbial dynamics correlate with therapeutic outcomes.

Participants were randomized into two groups: the SRP group (mechanical debridement only) and the Nd group (mechanical debridement with Nd:YAG laser therapy). Clinical parameters-including probing depth (PD), clinical attachment level (CAL), and gingival index (GI)-were assessed at baseline and 3 months post-treatment. Subgingival plaque samples were analyzed via 16S rDNA sequencing to characterize microbial community shifts.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-80 years
* Minimum of 14 remaining natural teeth
* Diagnosis of Stage III-IV periodontitis according to the 2018 World Workshop classification system
* No periodontal treatment within the past 6 months
* Willing to provide informed consent and participate in the study protocol

Exclusion Criteria:

* Presence of systemic conditions that may affect periodontal treatment outcomes (e.g., uncontrolled hypertension [>140/90 mmHg], diabetes mellitus [HbA1c >7%])
* Use of antibiotics or medications known to induce gingival enlargement (e.g., calcium channel blockers, phenytoin) within the past 3 months
* Coagulation disorders or hematologic diseases
* Active systemic infections
* Pregnancy or lactation
* Acute periodontal lesions
* Inability to comply with study protocols

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2024-08-28 (Actual); Primary Completion 2025-03-20 (Actual); Study Completion 2025-07-24 (Estimated)

PRIMARY OUTCOMES:
Alpha diversity of subgingival microbiota | From enrollment to the end of treatment at 3 months
  The higher the alpha diversity, the greater the species richness and evenness of the microbial community.
Probing Depth | From enrollment to the end of treatment at 3 months
  Probing depth (PD) measures the distance from the gingival margin to the base of the periodontal pocket, clinically assessing periodontal attachment loss and tissue destruction.

SECONDARY OUTCOMES:
Beta diversity of subgingival microbiota | From enrollment to the end of treatment at 3 months
  Beta diversity reflects the similarity in species composition.
Composition of subgingival microbiota | From enrollment to the end of treatment at 3 months
  The composition of subgingival microbiota refers to the taxonomic structure and relative abundance of bacterial species within the periodontal pocket biofilm, which plays a critical role in periodontal health and disease progression.
Microbial phenotypes of subgingival microbiota | From enrollment to the end of treatment at 3 months
  The microbial phenotypes of subgingival microbiota encompass the functional and metabolic characteristics of periodontal biofilm communities, including virulence factors, antibiotic resistance profiles, and synergistic interactions that contribute to periodontal pathogenesis.
Clinical Attachment Level (CAL) | From enrollment to the end of treatment at 3 months
  Clinical Attachment Level (CAL) measures the distance from the cementoenamel junction (CEJ) to the base of the periodontal pocket, directly quantifying periodontal tissue destruction and tooth-supporting structure loss.
Gingival Index (GI) | From enrollment to the end of treatment at 3 months
  The Gingival Index (GI) assesses the severity of gingival inflammation through standardized scoring of redness, swelling, and bleeding tendency, providing a quantitative measure of periodontal tissue health.
Plaque Index (PI) | From enrollment to the end of treatment at 3 months
  The Plaque Index (PI) quantifies the extent of bacterial plaque accumulation on tooth surfaces, using standardized scoring systems to assess oral hygiene status and periodontal disease risk.
Bleeding on Probing (BOP) | From enrollment to the end of treatment at 3 months
  Bleeding on Probing (BOP) evaluates gingival inflammation by recording the presence/absence of bleeding within 30 seconds after gentle periodontal probing, serving as a key diagnostic indicator of active periodontal disease.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China

DOCUMENTS (2):
  • Study Protocol (2024-08-16): https://cdn.clinicaltrials.gov/large-docs/56/NCT07061756/Prot_000.pdf
  • Informed Consent Form (2024-08-16): https://cdn.clinicaltrials.gov/large-docs/56/NCT07061756/ICF_001.pdf